CLINICAL TRIAL: NCT06734663
Title: Clinical Outcomes of Sutured Versus Sutureless Conjunctival Autograft in Primary Pterygium Excision
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amal Sherif Sayed Abdelrehim, Resident at Ophthalmology department, Faculty of medicine, Assiut University, Assiut University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB
Record Dates: First submitted 2024-11-17; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Pterygium of Conjunctiva and Cornea; Pterygium of Both Eyes; Pterygium
Keywords: pterygium surgery; sutureless pterygium; autologous blood; serum; pterygium excision using autologous blood in comparison to using sutures; new techniques in pterygium surgery
MeSH Terms: conditions — Pterygium Of Conjunctiva And Cornea; Pterygium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- pterygium excision using sutured technique (Placebo Comparator): This represents the main used technique in pterygium surgery that we will compare the less familiar sutureless technique to. pterygium is surgically removed and conjuctival graft is placed using sutures
  Interventions: Procedure: Clinical outcomes of sutured versus sutureless conjunctival autograft in primary pterygium excision; Procedure: pterygium excision and conjuctival graft suturing
- sutureless technique (Active Comparator): this represents the experimented technique in which pterygium excision is done and the graft is placed sutureless.
  Interventions: Procedure: Clinical outcomes of sutured versus sutureless conjunctival autograft in primary pterygium excision; Procedure: pterygium excision and conjuctival graft placement by autologous blood

INTERVENTIONS:
Procedure: Clinical outcomes of sutured versus sutureless conjunctival autograft in primary pterygium excision — Studies have concluded that pterygium surgical excision is the main treatment for pterygium. Pterygium excision with superior graft is the procedure followed most commonly at present. This is achieved by many methods, with the result differing from one method to another. The most important difference is the incidence of recurrence(4)But Varioustechniques such as Bare Sclera, Rotational Conjunctival Flap, Limbal Conjunctival Autograft, Amniotic Membrane Graft, and Free Conjunctival Autograft are also used for the removal of pterygium(3 ,4)Of the various possible alternative approaches, conjunctival autograft is usually preferred. Diverse methods for grafting with sutures, glue or autologous serum from the recipient bed are in use (5,6). Many adjunctive therapies like mitomycin C, corticosteroids, thiotepa, interferon-alpha- 2b, beta irradiation, 5-FU are being used to decrease the risk of recurrence after surgical removal of pterygium.
Procedure: pterygium excision and conjuctival graft suturing — pterygium is surgically removed, and a conjuctival graft is placed on bare sclera using sutures to surrounding conjuctiva.
  Arms: pterygium excision using sutured technique
Procedure: pterygium excision and conjuctival graft placement by autologous blood — pterygium is surgically removed and a conjuctival graft is placed on bare sclera on which the patient's blood remains. the graft is left without sutures, adhering only by autologous blood.
  Arms: sutureless technique

SUMMARY:
The goal of this study is to find out if a certain technique in pterygium excision surgery ,using no sutures, is better than the technique mostly used ,which uses sutures.

Investigators aim to find out whether the no sutures technique provides better efficiency and patient satisfaction than the traditional approach. They predict that if this study provides evidence of the advantages of this technique over the one used, surgeons would be encouraged to use it instead. Because not only would the patient benefit, the surgeon also may save operative time and effort used in the technique which uses sutures.

DETAILED DESCRIPTION:
This study is a comparative interventional study, in which patients are assigned into two groups comparable in age, gender, and general condition. The first group consists of patients with primary pterygium who will undergo surgery in a traditional approach in which the pterygium is surgically removed and after which a conjuctival graft is placed on the exposed sclera and sutured to the surrounding conjuctiva; in comparison, patients of the second group undergo pterygium excision in a similar matter initially.But the conjuctival graft is placed on the exposed sclera without suturing it to the nearby conjuctiva; instead, the graft remains in place using the patient's autologous blood. Fresh blood is left under the graft, while the surgeon merely compresses the graft for a few minutes. The aim of this study is to reach a conclusion as to which technique is more beneficial, to the patient and surgeon.

Patients included in this study must have primary pterygium, no known hematological condition, and full consent to the study. Surgery time is recorded to compare the effect of avoiding sutures on the surgeon's speed. After that, Patients are followed up in documented certain intervals post-operative, to assess graft displacement, signs of inflammation, signs of bleeding under graft, and patients' overall discomfort and satisfaction.

Finally, the two groups are compared with all factors taken into consideration. The ultimate target is to document evidence of the efficiency of the sutureless technique and endorse its application by Ophthalmologists elsewhere.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18-60 years old.
* Patients diagnosed with primary Pterygium (Grades 1-4)

Exclusion Criteria:

* Patients unable to offer viable consent
* Patients with other significant ocular surface diseases, bleeding disorders, or systemic conditions affecting wound healing.)
* Recurrent pterygium
* Combined ocular surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-04-20 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
to evaluate the rate of conjuctival graft displacement in pterygium excision and graft placement without sutures | 3 months
  the most valuable aim in this comparative study is to document if the graft placed sutureless will remain in place.So, in each follow-up, graft is assessed in regards to placement.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Ophthalmology department Assiut university, Asyut, Asyut Governorate
  - Ophthalmology department, Assiut University hospital, Asyut

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol